CLINICAL TRIAL: NCT03197415
Title: Intradiscal Injection of Platelet-rich Plasma for Discogenic Pain in L-spine
Brief Title: Platelet-rich Plasma for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pei-Yuan Lee, MD (Other)
Collaborators: Aeon Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pei-Yuan Lee, MD, Superintendent, Show Chwan Memorial Hospital
Organization: Show Chwan Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-16025-RD-105064
Record Dates: First submitted 2017-04-13; First posted 2017-06-23 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Discogenic Pain; Platelet-rich Plasma
Keywords: Platelet-rich plasma; Intervertebral Disc Degeneration; Low Back Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP group (Experimental): Intradisc injection of autologous platelet-rich plasma gel
  Interventions: Other: Platelet-rich plasma

INTERVENTIONS:
Other: Platelet-rich plasma — intradiscal injection of plasma-rich platelet

SUMMARY:
This study aims to evaluate the effect of platelet-rich plasma (PRP) on discogenic low back pain by comparing the pre- and post-interventional outcomes in patients receiving intradiscal injection of autologous PRP.

DETAILED DESCRIPTION:
Intervertebral disc (IVD) degeneration is an important clinical problem that often contributes to low back pain and degenerative disc diseases. Degeneration of the IVD induces anulus tears and fissures, which can cause severe discogenic low back pain. Because the IVD has little potential to self-regenerate, treatment of degenerative disc disease is one of the most challenging clinical problems facing the spine surgeon. Platelet-rich plasma (PRP) is a fraction of plasma that contains platelets and multiple growth factors concentrated at high level. Because activated platelets have the potential to release growth factors, PRP has been clinically used to accelerate wound healing and tissue regeneration in orthopedic and oral surgery. The soluble releasate isolated from PRP has recently been demonstrated to influence the metabolism of intervertebral discs in vitro. Furthermore, an intradiscal injection of autologous PRP has been shown to induce restoration of structural changes in the rabbit annular injection model in vivo. This clinical trial aims to investigate the safety and efficacy of intradiscal PRP injection in patients with discogenic low back pain. The pre- and post-interventional imaging and clinical outcomes will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years
* L-spine disc degeneration diagnosed by MRI
* Low back pain

Exclusion Criteria:

* Herniated disc
* With prior history of spine surgery
* With current or prior history of cancer
* With current or prior history of hematological disease
* Pregnancy
* Patients who will not cooperate with one-year followup

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
1-month postoperative function evaluated by Oswestry Disability Index | 1-month postoperative
  Function is evaluated using Oswestry Disability Index.

SECONDARY OUTCOMES:
4-month postoperative function evaluated by Oswestry Disability Index | 4-month postoperative
  Function is evaluated using Oswestry Disability Index
1-month postoperative pain evaluated by visual analogue scale | 1-month postoperative
  Pain is evaluated using visual analogue scale
4-month postoperative pain evaluated by visual analogue scale | 4-month postoperative
  Pain is evaluated using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, Study Chair — Show Chwan Memorial Hospital
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No